CLINICAL TRIAL: NCT05563155
Title: Repeat Dose Steroid to Prevent Pain Relapse After Total Knee Arthroplasty in Patients With High Pain Response - A Randomized Double-blind Placebo-controlled Trial
Brief Title: Repeat Dose Steroid to Prevent Pain Relapse After Total Knee Arthroplasty in Patients With High Pain Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Repeat Dose
Record Dates: First submitted 2022-09-16; First posted 2022-10-03 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Post Operative Pain, Acute
Keywords: Dexamethason; repeat; glucocorticoids; TKA surgery; steroids; High Pain Responders; postoperative pain; repeat dosing; FAST-TRACK
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: A double-blind randomization will be carried out, 5:5 block-randomization, half of which will be allocated to the CG and the other half to RDG.
  Group 1: Postoperative placebo tablet on day 1 after surgery.
  Group 2: Postoperative dexamethasone 24 mg tablet on day 1 after surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding The patient, all personnel attending in treatment and care of the patient, the investigators and the sponsor will all be blinded to the study-drug allocation, until all data processing is finished.
  The randomization-sequence will be stored in a sealed envelope at the Pharmacy at Lillebaelt Hospital who carried out the packaging-process. The randomization personnel have no contact to the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo tablet on day 1 after surgery given as one single dose. (Placebo Comparator): Control Group (CG):
  Intervention: Postoperative oral placebo tablet on day 1 after surgery given as one single dose.
  Interventions: Drug: Placebo
- Dexamethasone 24 mg on day 1 after surgery given as one single dose. (Active Comparator): Repeat Dose Group (RDG):
  Intervention: Postoperative oral dexamethasone 24 mg on day 1 after surgery given as one single dose.
  Interventions: Drug: Dexamethasone 24 mg

INTERVENTIONS:
Drug: Dexamethasone 24 mg — Dexamethasone 24 mg on day 1 after surgery.
  Other Names: Dexa-ratiopharm
  Arms: Dexamethasone 24 mg on day 1 after surgery given as one single dose.
Drug: Placebo — Placebo tablet given on day 1 after surgery.
  Arms: Placebo tablet on day 1 after surgery given as one single dose.

SUMMARY:
The aim of the study is to compare the effect of a repeat moderate dose of glucocorticoids postoperatively after preoperative high dose upon postoperative pain after Total Knee Arthroplasty (TKA) in an High Pain Respondes (HPR) population to a standard single high dose systemic preoperative administration in an HPR population.

As a standard procedure, all patients referred to the outpatient clinic due to suspected degenerative knee disease will be asked to fulfill the Pain Catastrophizing Scale (PCS). If TKA is decided, patients with a PCS score above 20 will be treated with intravenously administered Dexamethasone 1 mg/kg as a rounded-up-dose to closest 10 mg according to our guideline for FAST-TRACK TKA.

The repeat-dosing group (RDG) will receive a dose of 24 mg dexamethasone tablets at 9-11 pm on the first postoperative day. The control-group (CG) will receive placebo tablets at 9-11 pm on the first postoperative day.

DETAILED DESCRIPTION:
Total hip and knee arthroplasty (THA/TKA) are frequently performed procedures and are expected to increase in numbers along with the growing elderly population the next decade.

Total Knee Arthroplasty (TKA) is suitable for FAST-TRACK surgery, and is often performed as outpatient surgery with no hospital overnight stay.

Challenges in FAST-TRACK surgery include postoperative pain, nausea and vomiting (PONV), complications due to rescue-analgesics and surgical complications.

Pain is a well-known clinical problem, with up to 75% of TKA patients experiencing moderate to severe pain the first day after surgery, and 30-40% still experiencing moderate to severe pain 2 weeks after surgery, potentially delaying ambulation and recovery within the first weeks.

The role of severe acute postoperative pain upon the development of chronic pain is debatable, but important.

Data from our recently finished study in High Pain Responders (HPR), defined as patients with a score above 20 on the Pain Catastrophizing Scale (PCS), receiving preoperative high dose dexamethasone (Nielsen et al.: IN PREPARATION, clinicaltrials.gov ID NCT03763734, EudraCT 2018-002635-23, VEK H-18034778) found a persistent moderate to severe pain in 40 % of patients, at time 48 hours after surgery, corresponding to the time when the physiological effect of our dexamethasone intervention declines.

Moderate to severe pain (Visual analogue scale (VAS >30)) 24 hours postoperatively during a 5-meter walk test was associated with relapse pain at 48 hours.

Other studies have made attempts of investigating the effect of a repeated dose of steroids after TKA and Total Hip Arthroplasty (THA), but all have done so with a postoperative injection of low dose steroids. No previous studies have, to our knowledge, investigated the effects of repeat dosing after a preoperative high dose of steroid, and none focused on patients selected by their postoperative pain response. In spite of many studies and systematic reviews on the subject, the optimal timing and dose for steroid-intervention in TKA in different patient groups is still inadequately understood

The study conduct with a repeat moderate dose of steroids given as an oral tablet at 9-11 pm on the day after TKA surgery in patients receiving preoperative high dose steroids, who have a high postoperative pain response, in a FAST-TRACK perioperative setting. Oral administration of the repeat dose will allow for possible early discharge in future clinical settings.

The hypothesis is that a repeat moderate dose of glucocorticoid will reduce the postoperative pain on postoperative day 2 and cumulated pain day 2-3 after TKA surgery, when compared to single high dose preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years.
* Primary unilateral TKA.
* Ability to participate in the study (understand written and spoken Danish language, self-reported pain and satisfaction).
* Signed written informed consent form.
* PCS >20.
* Moderate to severe postoperative pain (VAS >30) in a 5-meter walk test 22-26 hours after end of surgery.

Exclusion Criteria:

* Ongoing treatment of systemic glucocorticoids or other immunosuppressant treatment apart from inhaled steroids.
* Insulin-dependent diabetes.
* Pregnancy or breastfeeding.*
* Allergies concerning the study-drug.
* Mental disability that could impair a patient's decision-making capability of giving informed consent and not enabling valid data collection.
* Patients with known diagnoses of schizophrenia, ongoing psychosis, bipolar disease and/or a history of ongoing anti-psychotic treatment.
* Patients with modulated pain-reception (experience) based on other diseases or injuries, e.g. spinal cord or brain injury, severe polyneuropathies or neurologic disorders.
* Peripheral nerve block per- or postoperatively.

  * Pregnancy: No women with suspected or proven pregnancy are eligible for inclusion. The following will be considered as safe contraception: intrauterine device or hormonal contraception. For women aged between 40-50 years, a urine HCG test for pregnancy will be performed.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Postoperative pain after 48 hours / day 2 morning, according to VAS-scale | Day 2 morning
  The amount of patients with moderate postoperative pain in a 5 meter walk test day 2 morgning(48 hours) postoperatively after total knee-arthroplasty.
  Pain is monitored by the Visual Analog Scale(VAS) 0-100 mm, where 0 is no pain and 100 mm is the worst pain. Moderate pain is considered a VAS >30 mm.

SECONDARY OUTCOMES:
Cumulated pain upon ambulation, according to VAS-scale (0-100mm), in a 5-meter walk test | From day 2-3
  Pain is monitored by the Visual Analog Scale(VAS) 0-100 mm, where 0 is no pain and 100 mm is the worst pain. Moderate pain is considered a VAS >30 mm
Cumulated pain score, according to VAS-scale (0-100mm), at rest, upon ambulation in a 5-meter walk test and at night according to VAS-scale(0-100mm) | From day 2-7
  Pain is monitored by the Visual Analog Scale(VAS) 0-100 mm, where 0 is no pain and 100 mm is the worst pain. Moderate pain is considered a VAS >30 mm
Quality of sleep, lethargy, dizziness, and nausea postoperative registration, according to the VAS-scale(0-100mm) | From day 2-7
  ain is monitored by the Visual Analog Scale(VAS) 0-100 mm, where 0 is no pain and 100 mm is the worst pain. Moderate pain is considered a VAS >30 mm
Cumulative use of rescue analgesics per day. | From day 2-7
Patient satisfaction with analgesic regimen in a ordinal scale from 0 to 10 | Day 7
Number of re-admissions within 30 days, and reasons why (follow-up by EPJ on postoperative day 30) | Day 30
Morbidity and mortality (30-day follow-up by EPJ or telephone). | Day 30
  Number of participant with morbidity and mortality in the first 30 days. Follow-up by EPJ or telephone.
Why still in hospital, an audit into the reasons the patient has not yet been discharged from the ward | Day 7
  An investigation into reason of why our patients remain in the hospital in the days after total Knee Arthroplasty in our Fast-Track center. This is investigated through a questionnaire previously used in a similar investigation in our center.
  The questionnaire is filled in by our project nurse. the questionnaire is a checkmark schedule with predetermined reasons to stay in hospital like low bloodpressure, sedation, dizzyness, lack of physiotherapy and medical and surgical complications.
  The outcome assesment will be descriptive.

CONTACTS AND LOCATIONS:
Locations (1):
- Vejle Hospital. Orthopedic Surgery Department. Clinical Research Unit, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Yes The individual patient data will be made available in anonymized form.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available from the date of publication

REFERENCES:
- [Background] Pabinger C, Lothaller H, Portner N, Geissler A. Projections of hip arthroplasty in OECD countries up to 2050. Hip Int. 2018 Sep;28(5):498-506. doi: 10.1177/1120700018757940. Epub 2018 May 21. PMID 29783896
- [Background] Erivan R, Villatte G, Dartus J, Reina N, Descamps S, Boisgard S. Progression and projection for hip surgery in France, 2008-2070: Epidemiologic study with trend and projection analysis. Orthop Traumatol Surg Res. 2019 Nov;105(7):1227-1235. doi: 10.1016/j.otsr.2019.07.021. Epub 2019 Oct 9. PMID 31606338
- [Background] Romanini E, Decarolis F, Luzi I, Zanoli G, Venosa M, Laricchiuta P, Carrani E, Torre M. Total knee arthroplasty in Italy: reflections from the last fifteen years and projections for the next thirty. Int Orthop. 2019 Jan;43(1):133-138. doi: 10.1007/s00264-018-4165-7. Epub 2018 Oct 6. PMID 30293141
- [Background] Sloan M, Premkumar A, Sheth NP. Projected Volume of Primary Total Joint Arthroplasty in the U.S., 2014 to 2030. J Bone Joint Surg Am. 2018 Sep 5;100(17):1455-1460. doi: 10.2106/JBJS.17.01617. PMID 30180053
- [Background] Gromov K, Kjaersgaard-Andersen P, Revald P, Kehlet H, Husted H. Feasibility of outpatient total hip and knee arthroplasty in unselected patients. Acta Orthop. 2017 Oct;88(5):516-521. doi: 10.1080/17453674.2017.1314158. Epub 2017 Apr 20. PMID 28426262
- [Background] Chan EY, Blyth FM, Nairn L, Fransen M. Acute postoperative pain following hospital discharge after total knee arthroplasty. Osteoarthritis Cartilage. 2013 Sep;21(9):1257-63. doi: 10.1016/j.joca.2013.06.011. PMID 23973139
- [Background] Andersen LO, Gaarn-Larsen L, Kristensen BB, Husted H, Otte KS, Kehlet H. Subacute pain and function after fast-track hip and knee arthroplasty. Anaesthesia. 2009 May;64(5):508-13. doi: 10.1111/j.1365-2044.2008.05831.x. PMID 19413820
- [Background] Lavand'homme P. Transition from acute to chronic pain after surgery. Pain. 2017 Apr;158 Suppl 1:S50-S54. doi: 10.1097/j.pain.0000000000000809. No abstract available. PMID 28134653
- [Background] Lavand'homme PM, Grosu I, France MN, Thienpont E. Pain trajectories identify patients at risk of persistent pain after knee arthroplasty: an observational study. Clin Orthop Relat Res. 2014 May;472(5):1409-15. doi: 10.1007/s11999-013-3389-5. PMID 24258688
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Sullivan M, Bishop S, Pivik J. The pain catastrophizing scale: development and validation. Psychol Assess 1995; 7: 524-32
- [Background] Khan RS, Ahmed K, Blakeway E, Skapinakis P, Nihoyannopoulos L, Macleod K, Sevdalis N, Ashrafian H, Platt M, Darzi A, Athanasiou T. Catastrophizing: a predictive factor for postoperative pain. Am J Surg. 2011 Jan;201(1):122-31. doi: 10.1016/j.amjsurg.2010.02.007. Epub 2010 Sep 15. PMID 20832052
- [Background] Xu H, Zhang S, Xie J, Lei Y, Cao G, Pei F. Multiple Doses of Perioperative Dexamethasone Further Improve Clinical Outcomes After Total Knee Arthroplasty: A Prospective, Randomized, Controlled Study. J Arthroplasty. 2018 Nov;33(11):3448-3454. doi: 10.1016/j.arth.2018.06.031. Epub 2018 Jul 4. PMID 30033064
- [Background] Li D, Zhao J, Yang Z, Kang P, Shen B, Pei F. Multiple Low Doses of Intravenous Corticosteroids to Improve Early Rehabilitation in Total Knee Arthroplasty: A Randomized Clinical Trial. J Knee Surg. 2019 Feb;32(2):171-179. doi: 10.1055/s-0038-1636506. Epub 2018 Mar 7. PMID 29514368
- [Background] Xu B, Ma J, Huang Q, Huang ZY, Zhang SY, Pei FX. Two doses of low-dose perioperative dexamethasone improve the clinical outcome after total knee arthroplasty: a randomized controlled study. Knee Surg Sports Traumatol Arthrosc. 2018 May;26(5):1549-1556. doi: 10.1007/s00167-017-4506-x. Epub 2017 May 4. PMID 28474088
- [Background] Dissanayake R, Du HN, Robertson IK, Ogden K, Wiltshire K, Mulford JS. Does Dexamethasone Reduce Hospital Readiness for Discharge, Pain, Nausea, and Early Patient Satisfaction in Hip and Knee Arthroplasty? A Randomized, Controlled Trial. J Arthroplasty. 2018 Nov;33(11):3429-3436. doi: 10.1016/j.arth.2018.07.013. Epub 2018 Jul 19. PMID 30078660
- [Background] Kim JK, Ro DH, Lee HJ, Park JY, Han HS, Lee MC. Efficacy of Systemic Steroid Use Given One Day After Total Knee Arthroplasty for Pain and Nausea: A Randomized Controlled Study. J Arthroplasty. 2020 Jan;35(1):69-75. doi: 10.1016/j.arth.2019.08.026. Epub 2019 Aug 19. PMID 31563397
- [Background] Lei YT, Xu B, Xie XW, Xie JW, Huang Q, Pei FX. The efficacy and safety of two low-dose peri-operative dexamethasone on pain and recovery following total hip arthroplasty: a randomized controlled trial. Int Orthop. 2018 Mar;42(3):499-505. doi: 10.1007/s00264-017-3537-8. Epub 2017 Jun 25. PMID 28647788
- [Background] Lei Y, Huang Q, Xu B, Zhang S, Cao G, Pei F. Multiple Low-Dose Dexamethasone Further Improves Clinical Outcomes Following Total Hip Arthroplasty. J Arthroplasty. 2018 May;33(5):1426-1431. doi: 10.1016/j.arth.2017.11.057. Epub 2017 Dec 5. PMID 29258763
- [Background] Kehlet H, Joshi GP. The systematic review/meta-analysis epidemic: a tale of glucocorticoid therapy in total knee arthroplasty. Anaesthesia. 2020 Jul;75(7):856-860. doi: 10.1111/anae.14946. Epub 2019 Dec 4. No abstract available. PMID 31802486
- [Background] Riddle DL, Wade JB, Jiranek WA, Kong X. Preoperative pain catastrophizing predicts pain outcome after knee arthroplasty. Clin Orthop Relat Res. 2010 Mar;468(3):798-806. doi: 10.1007/s11999-009-0963-y. Epub 2009 Jul 8. PMID 19585177
- [Background] Toner AJ, Ganeshanathan V, Chan MT, Ho KM, Corcoran TB. Safety of Perioperative Glucocorticoids in Elective Noncardiac Surgery: A Systematic Review and Meta-analysis. Anesthesiology. 2017 Feb;126(2):234-248. doi: 10.1097/ALN.0000000000001466. PMID 27922839
- [Background] Jorgensen CC, Pitter FT, Kehlet H; Lundbeck Foundation Center for Fast-track Hip and Knee Replacement Collaborative Group. Safety aspects of preoperative high-dose glucocorticoid in primary total knee replacement. Br J Anaesth. 2017 Aug 1;119(2):267-275. doi: 10.1093/bja/aex190. PMID 28854533
- [Background] de la Motte L, Kehlet H, Vogt K, Nielsen CH, Groenvall JB, Nielsen HB, Andersen A, Schroeder TV, Lonn L. Preoperative methylprednisolone enhances recovery after endovascular aortic repair: a randomized, double-blind, placebo-controlled clinical trial. Ann Surg. 2014 Sep;260(3):540-8; discussion 548-9. doi: 10.1097/SLA.0000000000000895. PMID 25115430
- [Background] Carter R, Holiday DB, Grothues C, Nwasuruba C, Stocks J, Tiep B. Criterion validity of the Duke Activity Status Index for assessing functional capacity in patients with chronic obstructive pulmonary disease. J Cardiopulm Rehabil. 2002 Jul-Aug;22(4):298-308. doi: 10.1097/00008483-200207000-00014. PMID 12202852
- [Result] Rupp M, Lau E, Kurtz SM, Alt V. Projections of Primary TKA and THA in Germany From 2016 Through 2040. Clin Orthop Relat Res. 2020 Jul;478(7):1622-1633. doi: 10.1097/CORR.0000000000001214. PMID 32168057
- [Derived] Springborg AH, Varnum C, Nielsen NI, Rasmussen LE, Kjaersgaard-Andersen P, Pleckaitiene L, Gromov K, Troelsen A, Kehlet H, Foss NB. Repeat-dose dexamethasone to prevent pain relapse after total knee arthroplasty in high-pain-response patients: A randomised, double-blind, placebo-controlled superiority trial. Eur J Anaesthesiol. 2025 Jul 1;42(7):599-608. doi: 10.1097/EJA.0000000000002189. Epub 2025 May 14. PMID 40364780